CLINICAL TRIAL: NCT04057157
Title: Post-market Clinical Data Collection Plan for the Biodesign® Dural and Duraplasty Grafts
Brief Title: Post-market Assessment of Biodesign Dural Repair Grafts
Status: Completed | Type: Observational
Sponsor: Cook Research Incorporated (Industry)
Responsible Party: Sponsor
Organization: Cook Group Incorporated (Industry)
Other Study IDs: 17-10
Record Dates: First submitted 2019-08-13; First posted 2019-08-15 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Cerebrospinal Fluid Leak
Keywords: dura mater repair; cerebrospinal fluid leak; CSF leak; Biodesign® Dural Repair Graft; Biodesign® Duraplasty Repair Graft
MeSH Terms: conditions — Cerebrospinal Fluid Leak; Cerebrospinal Fluid Otorrhea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Device: Biodesign Dural or Duraplasty Repair Grafts — Patients will receive the Biodesign Dural or Duraplasty Repair Grafts according to the Instruction for Use.

SUMMARY:
The purpose of this clinical study is to gather post-market clinical evidence on the use of the Biodesign® Dural and Duraplasty Grafts when used as a dura substitute of the dura mater.

ELIGIBILITY:
Inclusion Criteria:

1. Planned use of the Biodesign Dural or Duraplasty Graft.

Exclusion Criteria:

1. Age <18 years
2. Unable or unwilling to provide informed consent
3. Life expectancy <6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have had dura mater repair using a Biodesign Dural or Duraplasty Graft.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Percentage of patients without clinically relevant cerebrospinal fluid (CSF) leakage | 2 months
  Clinically relevant CSF leakage is when it requires treatment (e.g., lumbar drain or surgical repair) or leads to an infection of the central nervous system (e.g., meningitis).

CONTACTS AND LOCATIONS:
Locations (3):
- University of Alabama Birmingham Hospital, Birmingham, Alabama, United States
- Toronto Western Hospital, Toronto, Ontario, Canada
- Ospedale Bellaria-Bolonga, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Cook Research Incorporated (CRI) is fully committed to supporting the principles of responsible data sharing, including providing qualified scientific researchers access to deidentified, patient-level data from CRI clinical studies to conduct legitimate scientific research. Data underlying the results reported in this clinical study will be made available for request after final report has been distributed and ending 5 years after final report has been distributed. Interested researchers may review the "Cook Research Incorporated Policy on Access to Clinical Study Data" at https://www.cookresearchinc.com/extranet/data-access.html and submit a complete research proposal to request data access. Additional study documents (such as the study protocol) will be shared as needed if the data access request is granted. A data sharing agreement will be executed for access to deidentified patient-level data.